CLINICAL TRIAL: NCT05375253
Title: A Phase I Trial of Donor Enriched Activated NK (DEA-NK) Cell Infusion Post Haploidentical Stem Cell Transplant for Refractory Myeloid Malignancies
Brief Title: Donor Enriched Activated NK Cell Infusion Post Haploidentical Stem Cell Transplant for Refractory Myeloid Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI has left institution and is taking the study with him.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0158-22-FB
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Donor Enriched Activated NK Infusion (DEA-NK) (Experimental): Infusion of DEA-NK on day +7 post-transplant
  Interventions: Biological: Donor Enriched Activated Natural Killer Cell Infusion

INTERVENTIONS:
Biological: Donor Enriched Activated Natural Killer Cell Infusion — αβ TCR/CD19 depleted (DEA-NK) cells on day +7 post T-cell replete Haplo-Tx with PTCY

SUMMARY:
Patients with relapse refractory myeloid malignancies have no therapeutic options for long term remission. Some success has been achieved in treating patients with refractory relapsed acute myeloid leukemia (AML) in using haploidentical cytokine activated natural killer (NK) cell immunotherapy. This process infuses natural killer (NK) cells from a half- or partially-matched donor. These cells are a type of lymphocytes made by a person's immune system that are important for fighting infection and tumor cells and are modified with other immune system substances to be more effective. One limiting factor is the recovery of recipient's immune system rejecting the infused NK cells. The use of haploidentical activated NK cell therapy post-transplant is a possible option to create longer lived infused NK cells and support cancer fighting ability.

DETAILED DESCRIPTION:
Patients with relapse refractory myeloid malignancies [acute myeloid leukemia (AML) myelodysplastic (MDS)/myeloproliferative (MPD) disorders] have no therapeutic options for long term remission. Haploidentical cytokine activated natural killer (NK) cell immunotherapy has been used with some success in treating patients with refractory relapsed AML. One limiting factor to the in-vivo expansion of infused activated NK cells is the recovery of recipient's immune system rejecting the infused NK cells. The use of haploidentical activated NK cell therapy post haploidentical transplant is an attractive option to induce in-vivo persistence of the infused NK cells and support anti leukemic efficacy.

This is a pilot trial testing the feasibility, safety and immunologic effects of dose escalated donor enriched activated natural killer cell infusion (DEA-NK) on day +7 post haploidentical stem cell transplantation. Participants must be adult patients with relapse refractory AML, MDS, or MPD, available haploidentical related donor, and adequate organ functions to undergo stem cell transplant. Participants will be followed for 6 months and 1 year following transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign informed Consent
2. Age > 19 years and ≤ 70 years.
3. Deemed eligible for allogeneic stem cell transplantation with a minimum KPS of 70% (Appendix A).
4. Available HLA-haploidentical related donor as defined in section 5.2.1
5. Subjects with adequate organ functions as measured by:

   1. Cardiac: Left ventricular ejection fraction at rest must be >45%,
   2. Hepatic: Bilirubin < 2.5 mg/dL except for Gilbert syndrome; and ALT, AST, and Alkaline Phosphatase < 5 x ULN.
   3. Renal: GFR > 50 mL/min/1.73m2,
   4. Pulmonary: FEV 1, FVC, DLCO ion capacity) > 45% predicted (corrected for hemoglobin); or 02 saturation > 92% on room air.
6. Able to be off of corticosteroids (10 mg or less of prednisone or equivalent doses of other systemic steroids are allowed) and any other immune suppressive medications beginning on Day -3
7. Subjects with prior central nervous system (CNS) involvement are eligible provided that it has been treated and cerebral spinal fluid (CSF) is clear for at least 2 weeks prior to enrollment. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
8. Clinical diagnosis of one of the following:

A. Refractory AML without complete remission (CR) after 2 or more cycles of induction therapy (primary induction failure), or AML relapsed after obtaining a CR and failed one or more cycles of re-induction therapy. decitabine or azacytidine with venetoclax will be considered as one cycle of induction therapy.

B. Myelodysplastic Syndrome+/- myeloproliferative neoplasm MDS/MPN which failed to adequately respond (persistence of blasts >5%) to hypomethylating agents and or chemotherapy (minimum of 3 cycles of hypomethylating agents or 2 cycles of hypomethylating + venetoclax or one cycle of induction chemotherapy)

Exclusion Criteria:

1. Autologous hematopoietic stem cell transplant < 3 months prior to enrollment.
2. Circulating peripheral blood blast count > 1000/µl (despite hydroxyurea and or leukapheresis).
3. Previous allogeneic stem cell transplant.
4. Presence of donor specific antibodies (DSA) with Mean Fluorescence Intensity (MFI) of ≥5000 as assessed by the single antigen bead assay, < 6 weeks prior to starting transplant conditioning
5. Uncontrolled angina, severe uncontrolled ventricular arrhythmias.
6. Received any investigational drugs within the 14 days prior to the first day of transplant conditioning (starting on day -6)
7. Women of child-bearing potential must not be pregnant and/or breastfeeding

   a. Note: All females with intact ovaries and uterus will have two pregnancy tests as part of standard of care pre-transplant protocols.
8. Evidence of HIV infection or known HIV positive serology (completed as part of pre-transplant testing).
9. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
10. Non-hematologic malignancy within prior three (3) years, with the exception of squamous cell or basal cell skin carcinoma.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Percent of successful DEA-NK cell infusions | 100 Days
  Assess the feasibility of infusing activated enriched donor natural killer cell infusion (DEA-NK) at day +7 post-transplant by the ability to manufacture and administer the DEA-NK cells at study dose levels.
Number of adverse events for those who have a DEA-NK cell infusion | 100 Days
  Assess safety of the DEA-NK cell infusions by recording adverse events experienced by subjects at each dose level.
Maximum tolerated dose of DEA-NK cell infusions | 100 Days
  To determine the maximum tolerated dose (MTD) of DEA-NK cell infusion as determined by dose limiting toxicities (DLT) observed.

SECONDARY OUTCOMES:
Non-Relapse Mortality Rate | 1 year
  Non-Relapse Mortality (NRM) at 100 days, 180 days and 1 year
Time to neutrophil recovery | 21 Days
  Time to neutrophil recovery defined as the first of 3 consecutive days following the nadir that the absolute neutrophil count is at least 500/µl
Time to platelet recovery | 21 Days
  Time to platelet recovery defined as the first day that the platelet count is at least 20,000/µl without a transfusion in the preceding 7 days
Incidence of graft failure | 35 Days
  Incidence of graft failure as defined by ANC < 500/µl by Day +35 in the absence of disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No